CLINICAL TRIAL: NCT00901992
Title: Evaluation of a Self-management Oriented Diabetes Education Program for the Initiation of Intensive Insulin Therapy in Type 2 Diabetic Patients
Brief Title: Evaluation of a Self-management Oriented Diabetes Education Program for Intensified Insulin Therapy in Type 2 Diabetes
Acronym: MEDIAS-2-ICT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Forschungsinstitut der Diabetes Akademie Mergentheim (Other)
Responsible Party: Principal Investigator, Norbert Hermanns, Prof. Dr., Forschungsinstitut der Diabetes Akademie Mergentheim
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FIDAM-02-09
Record Dates: First submitted 2009-05-12; First posted 2009-05-14 (Estimated); Last update posted 2014-08-11 (Estimated); Status verified 2014-08

CONDITIONS: Type 2 Diabetes
Keywords: type 2 diabetes; education; self-management; insulin therapy
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- MEDIAS 2 ICT (Experimental): MEDIAS 2 ICT - education program for the initiation of intensive conventional insulin treatment (ICT) in type 2 diabetic patients
  Interventions: Behavioral: MEDIAS 2 ICT
- Current ICT program (ACC) (Active Comparator): This education program consists of 10 lessons combining an insulin education program with an hypertension program
  Interventions: Behavioral: Current ICT program (ACC-ICT)

INTERVENTIONS:
Behavioral: MEDIAS 2 ICT — MEDIAS 2 ICT is a newly developed education program for the initiation of intensive conventional insulin therapy in type 2 diabetic patients (10 lessons of group sessions for 4-8 participants)
  Arms: MEDIAS 2 ICT
Behavioral: Current ICT program (ACC-ICT) — This program is conducted in 10 lessons in a group setting (4-8 participants)
  Arms: Current ICT program (ACC)

SUMMARY:
A new diabetes education program for the initiation of intensive insulin therapy in type 2 diabetic patients (MEDIAS 2 ICT) was developed.

In the evaluation, this new developed program is compared with an education programs which is currently used for diabetes education. It is expected that the new developed program (MEDIAS 2 ICT) can demonstrate non-inferiority with regard to the main outcome variable glycemic control. If non-inferiority can be demonstrated superiority of this programs will be tested.

The results regarding the intervention arms "MEDIAS ICT" vs. " ACC" (control condition) will be separately analyzed and published.

DETAILED DESCRIPTION:
The MEDIAS 2 ICT program is based on a self-management/empowerment approach. It is conducted as a group program comprising 10 lessons of 90 minutes each. MEDIAS 2 ICT is designed to help patients perform multiple-injection insulin therapy and adjust their insulin doses depending on carbohydrate consumption, physical exercise, and pre-prandial glucose levels. In addition, MEDIAS 2 ICT focuses on controlling metabolic risk factors (elevated lipids and blood pressure), coping with the risk of late complications, and reducing the emotional burden of diabetes and its treatment.

The active comparator condition (ACC) consist of a combination of two previously established and evaluated education programs - a diabetes education program to initiate mealtime insulin and a hypertension education program for the treatment of hypertension. These education programs were developed in the 1980s and 1990s and were more didactic-oriented, focusing primarily on the acquisition of knowledge, skills, and information about the correct treatment of diabetes and hypertension.

Both treatment arms (MEDIAS 2 ICT and ACC) consisted of 10 lessons, which were conducted as group sessions.

ELIGIBILITY:
Inclusion Criteria:

* type 2 diabetes
* age < 75 and age > 17 years
* two years diabetes duration with oral treatment
* BMI > 20 nad BMI < 40 kg/m²
* informed consent

Exclusion Criteria:

* current psychiatric disease
* dementia or other severe cognitive impairment
* severe complications
* severe conditions (e.g., cancer)
* gestational diabetes

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 186 (Actual)
Dates: Start 2009-05; Primary Completion 2010-04 (Actual); Study Completion 2010-08 (Actual)

PRIMARY OUTCOMES:
A1c values | six month follow up after termination of the programs

SECONDARY OUTCOMES:
Quality of life using the SF 12 mental and physical composite scales | six month follow up
diabetes knowledge (Diabetes knowledge test for insulin treatment in type 2 diabetes) | 6 month follow up
diabetes related distress (Problem areas in Diabetes Questionnaire -PAID) and satisfaction with insulin therapy (Insulin Treatment Experience Questionnaire ITEQ) | 6 month follow up
Self care behavior (Summary of Self-Care Activities Scale) | 6 month follow up
lipids (total cholesterol, triglycerides, HDL and LDL) | 6 month follow up
weight (Body mass index) | 6 month follow up

CONTACTS AND LOCATIONS:
Overall Officials: Norbert Hermanns, PhD, Principal Investigator — Forschungsinstitut der Diabetes Akademie Mergentheim
Locations (1):
- Diabetes Centre Mergentheim, Bad Mergentheim, Germany

REFERENCES:
- [Result] Hermanns N, Kulzer B, Maier B, Mahr M, Haak T. The effect of an education programme (MEDIAS 2 ICT) involving intensive insulin treatment for people with type 2 diabetes. Patient Educ Couns. 2012 Feb;86(2):226-32. doi: 10.1016/j.pec.2011.05.017. Epub 2011 Jun 28. PMID 21715124